CLINICAL TRIAL: NCT00502970
Title: A Randomized Trial Comparing a Short Course Versus Standard Treatment in Patients With Chronic Hepatitis C Virus Infection
Brief Title: Short Course of Interferon Treatment in Patients With HCV Infection
Acronym: STAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Getz Pharma (Industry)
Responsible Party: Proffessor Saeed Hamid, The Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 302-Med/ERC-04
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Hepatitis C; Chronic Disease; Treatment
Keywords: Chronic HCV; Treatment
MeSH Terms: conditions — Hepatitis C; Chronic Disease | interventions — Ribavirin; Iron-Dextran Complex; Interferons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 16 weeks Interferon Tiw with Ribavirin
  Interventions: Drug: 16 weeks Interferon Tiw with Ribavirin
- 2 (Active Comparator): 24 weeks Interferon Tiw with Ribavirin
  Interventions: Drug: 24 weeks Interferon

INTERVENTIONS:
Drug: 16 weeks Interferon Tiw with Ribavirin — 16 weeks Interferon Tiw
  Other Names: Uniferon
  Arms: 1
Drug: 24 weeks Interferon — 24 weeks Interferon Tiw with Ribavirin
  Other Names: Uniferon
  Arms: 2

SUMMARY:
To determine if a shorter course of interferon and ribavirin therapy will be sufficient in carefully selected patients with chronic hepatitis C virus genotype 3 infection, as compared to the standard length of treatment of 6 months.

DETAILED DESCRIPTION:
1. INTRODUCTION

   1.1 Hepatitis C Hepatitis C Virus (HCV) is a major cause of chronic hepatitis and hepatic fibrosis1. Acute infection advances to chronicity in up to 80% of patients, which can further progress to cirrhosis and hepatocellular carcinoma in a significant number1.

   Hepatitis C is a global problem, prevalent in industrialized as well as in the developing world2. It is a major cause of chronic liver disease (CLD) in Pakistan and has surpassed hepatitis B as the single most important cause for cirrhosis and hepatocellular carcinoma (HCC) in Pakistan 3.

   1.2 Study Medications A combination of interferon and ribavirin therapy has been the standard of care world-wide for the past few years1, 2. Standard treatment duration is for 24 weeks for genotype non 1, and 48 weeks for genotype 12.

   1.2.1 Interferon Alfa 2a Interferon Alfa was the first drug shown to have bioactivity against HCV. Combining ribavirin with interferon Alfa was found to be more effective than interferon Alfa mono-therapy in previously untreated patients as well in patients who relapsed after one or more courses of interferon Alfa therapy2.

   1.2.2 Ribavirin Ribavirin is a guanosine analogue that inhibits the in vitro replication of a wide range of RNA and DNA viruses1. The mechanism of antiviral activity is not fully defined, although it may involve alteration of cellular nucleotide pools and inhibition of viral RNA synthesis1, 4. Ribavirin monotherapy has little or no effect on the replication of HCV but can result in normalization of serum ALT activity and improvement in liver histology. However, relapse occurs in nearly all patients treated with ribavirin alone1.

   Combining Ribavirin with Interferon has been found to be more effective than Interferon monotherapy in the treatment of chronic hepatitis C. In a large clinical trial of 1121 patients, a sustained virological response (SVR) was achieved in 53% of patients treated with Interferon plus Ribavirin as compared to 29% of patients treated with Interferon alone1, 4.
2. RATIONALE Most treatment related studies on HCV have come from the West, where the most prevalent genotype is 1; their results however do not necessarily reflect the outcome in a developing country like Pakistan, where studies have already confirmed that the most prevalent genotype is 32. Success rates have globally been reported to be high when treating genotype 3: it has long been observed that patients infected with genotype 2 and 3 respond better to interferon therapy than patients infected with genotype 11, 3.

   Favorable prognostic factors have been identified which predict a better response to therapy in the treatment of chronic HCV. These include:
   * Younger age
   * Genotype 3
   * No cirrhosis on liver biopsy, and
   * Absence of alcohol or drug abuse1, 7.

   Few studies have investigated the efficacy of a short course therapy for patients with favorable predictive factors; most of these studies have used interferon monotherapy4, 5, while others have used a combination treatment for shorter duration in relapsed patients6. There is evidence that combination treatment may be beneficial when used as induction therapy, followed by interferon in a short course program, 7. Cases infected with HCV genotype 3 being treated for as little as 4-12 weeks and remaining sustained responders have been reported8

   Since HCV genotype 3 responds so well to a combination of interferon and Ribavarin, it has been suggested that this patient population may have a similar response to a shorter duration of therapy7, 8, 9. The efficacy of a short course interferon and Ribavarin combination therapy compared to a longer course of therapy has not been compared in the treatment of patients with favorable predictive factors.

   2.1 Rationale for Dosage Selection

   1.2.2.1 Interferon Alfa 2a The dose chosen for interferon Alfa 2a (3 million units thrice weekly, sc) is the dose currently approved in Pakistan for combination therapy with ribavarin1.

   1.2.2.2 Ribavarin The dose chosen for Ribavarin (800-1200 mg per day) is the dose currently approved in Pakistan for combination therapy with interferon in patients with HCV.1
3. HYPOTHESIS In patients with chronic hepatitis C infection with favorable predictive factors for treatment, a short course of combination therapy with interferon and Ribavarin is equally efficacious as the longer course of treatment.
4. OBJECTIVE To determine whether 16 weeks of interferon and Ribavarin therapy is as effective as 24 weeks of therapy in achieving sustained virological response in patients with favorable predictive factors who are infected with HCV genotype 3.
5. SIGNIFICANCE Pakistan has an enormous burden of chronic HCV infection. The cost of treatment is prohibitive and is unaffordable for a large proportion of our population2, 3. A short course therapy comparable to the standard regimen would have significant implications; a striking decrease in financial burden on the health care system of the country, as well as the patients and a reduction in patient exposure to both medications, resulting in decreased treatment related adverse effects. In addition a larger number of patients will be able to afford the treatment due to a decrease in treatment duration and in turn the overall cost.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and non-pregnant females (more than 18 and less than equal to 50 years of age).
* Treatment naïve patients.
* Serological evidence of hepatitis C infection by an anti-HCV antibody test
* HCV PCR positive
* Genotype 3
* Absence of cirrhosis on liver biopsy.
* Absence of alcohol or drug abuse.

Exclusion Criteria:

* Patients who do not consent to be included in the study.
* Pregnant or breast feeding females.
* Patients with a hemoglobin of <10g/dl, ANC <1500c/mm, and a platelet count <90000c/mm.
* Genotype non 3
* HCV PCR positive at the end of 4 weeks of treatment.
* Presence of cirrhosis on liver biopsy.
* Decompensated liver disease.
* History or other evidence of a medical condition associated with chronic liver disease other than CHC (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposure)
* History of having received IFN, PEG-IFN, RBV therapy previously.
* History of systemic antiviral therapy or investigational drug 3 months prior to the first dose of study treatment.
* Patients expected to need systemic antiviral therapy at any time during their participation in the study.
* Exceptions from the last two exclusion criteria are patients who have had a limited (less than 7 day) course of acyclovir or valacyclovir for herpetic lesions more than 1 month prior to the first administration of trial treatment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2004-05; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Sustained Virological response | six months after stopping treatment

SECONDARY OUTCOMES:
Safety of short course of Interferon & Ribavirin | Four or Six months

CONTACTS AND LOCATIONS:
Overall Officials: Saeed S Hamid, FRCP, Principal Investigator — Aga Khan University
Locations (1):
- The Aga Khan University, Stadium Road, Karachi, Sindh, Pakistan